CLINICAL TRIAL: NCT05484154
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of 3K3A-APC in Combination with Tissue Plasminogen Activator, Mechanical Thrombectomy, or Both in Subjects with Moderate to Severe Acute Ischemic Stroke
Brief Title: Efficacy and Safety Evaluation of 3K3A-APC in Ischemic Stroke
Acronym: RHAPSODY-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: NIH funding suspension.
Sponsor: ZZ Biotech, LLC (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Southern California (Other); University of Cincinnati (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZZ-3K3A-301; UG3NS119199 (NIH)
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Stroke; APC; 3K3A; 3K3A-APC; Activated protein C; RHAPSODY
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — 3K3A-APC protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10mg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- 15mg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- 30mg of 3K3A-APC (Active Comparator): 3K3A-APC, q12h for up to 5 doses
  Interventions: Biological: 3K3A-APC
- Placebo (Placebo Comparator): Matching placebo, q12h for up to 5 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 3K3A-APC — 3K3A-APC, diluted in 0.9% sodium chloride in water, given at 100 mL IV infusion
  Other Names: 3K3A-Activated Protein C
  Arms: 10mg of 3K3A-APC; 15mg of 3K3A-APC; 30mg of 3K3A-APC
Other: Placebo — Matching placebo, 0.9% sodium chloride in water, given at 100 mL IV infusion
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravenous doses of 3K3A-APC, a recombinant variant of human activated protein C (APC), in the treatment of acute ischemic stroke following treatment with thrombolysis, mechanical thrombectomy or both.

DETAILED DESCRIPTION:
This multicenter, randomized, placebo-controlled, double-blind, Phase 3 study is being performed in coordination with StrokeNet to evaluate efficacy and safety of 3K3A-APC following administration of thrombolysis, mechanical thrombectomy, or both in subjects with moderate to severe acute ischemic stroke.

The study will be conducted in two phases. During a lead-in dose-finding phase, a maximum of 360 subjects will be randomized to 3K3A-APC or placebo using a Bayesian adaptive approach. Randomized subjects will receive 3K3A-APC or placebo every 12 hours for up to 5 doses (approximately 3 days) or until discharge from the hospital (whichever occurs first). The lead-in phase will transition to one selected 3K3A APC dose-and recruitment will continue-when a single dose proves superior to all other doses and safe.

The definitive phase will continue with the selected dose of 3K3A-APC from the lead-in phase. Randomization will be stratified on 4 variables. Lead-in patients who received the dose selected for the definitive phase will be included in the final data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Able to receive thrombolysis, mechanical thrombectomy or both
* National Institutes of Health Stroke Scale (NIHSS) score of ≥ 5
* Signed informed consent
* Agreement to use effective birth control throughout the study

Exclusion Criteria:

* Neurologic deficit is non-disabling
* History of stroke or penetrating head injury within 90 days prior to enrollment
* History of previous or current diagnosis of intracranial hemorrhage
* Moyamoya disease, cerebral arteriovenous malformation, or known unsecured aneurysm requiring intervention during the acute study period
* Presence of tandem lesions suggesting a likely need for proximal artery stenting during the thrombectomy procedure that would mandate post-operative dual antiplatelet therapy
* Presence of other neurological or non-neurological co-morbidities, independently of the current stroke, that may lead to further deterioration in the subject's neurological status during the study period
* Prolonged prothrombin time (PT) or activated partial thromboplastin time (aPTT)
* Severe hypertension or hypotension
* Blood glucose concentration < 50 mg/dL
* Prior exposure to any exogenous form of a recombinant variant of human APC

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of 3K3A-APC on 90-day disability | Day 90 mRS
  Day 90 mRS scores will be compared between groups using ordinal (shift) analysis

SECONDARY OUTCOMES:
To evaluate the safety of 3K3A-APC | Baseline to Day 90
  The percentage of subjects who experienced any treatment-related AE will be compared using a Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D Lyden, MD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No